CLINICAL TRIAL: NCT06698549
Title: A Phase 1 Non-Randomized, Open-Label, Multiple Dose Study to Evaluate the Pharmacokinetics, Safety and Tolerability of ALG-097558 in Subjects With Renal Impairment and in Healthy Subjects With Normal Renal Function
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety and Tolerability of ALG-097558 in Subjects With Renal Impairment and in Healthy Subjects With Normal Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aligos Therapeutics (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALG-097558-703 / DMID 24-0022
Record Dates: First submitted 2024-11-12; First posted 2024-11-21 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2024-11

CONDITIONS: COVID 19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This study is non-randomized, open-label, parallel group study. In Part 1, Cohort 1 will enroll severely renally impaired subjects and Cohort 2 will enroll subjects without renal impairment. In Part 2, if triggered, Cohort 3 will enroll mildly renally impaired subjects and Cohort 4 moderately renally impaired subjects. Cohort 5 will enroll subjects without renal impairment.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Subjects with Severe Renal Impairment (Experimental): Subjects with severe renal impairment will receive oral doses of 300 mg ALG-097558 twice daily (every 12 hours [Q12H]) for 6 days for 11 total doses.
  Interventions: Drug: ALG-097558
- Subjects with Normal Renal Function (Experimental): Subjects with normal renal function will receive oral doses of 300 mg ALG-097558 twice daily (every 12 hours [Q12H]) for 6 days for 11 total doses.
  Interventions: Drug: ALG-097558
- Subjects with Mild Renal Impairment (Optional) (Experimental): Subjects with mild renal impairment will receive oral doses of 300 mg ALG-097558 twice daily (every 12 hours [Q12H]) for 6 days for 11 total doses.
  Interventions: Drug: ALG-097558
- Subjects with Moderate Renal Impairment (Optional) (Experimental): Subjects with moderate renal impairment will receive oral doses of 300 mg ALG-097558 twice daily (every 12 hours [Q12H]) for 6 days for 11 total doses.
  Interventions: Drug: ALG-097558

INTERVENTIONS:
Drug: ALG-097558 — Multiple doses of ALG-097558 300 mg (3 x 100 mg tablets)

SUMMARY:
This is a Phase 1 non-randomized, open-label, multiple dose, parallel-group study of ALG-097558 in subjects with severe renal impairment and subjects without renal impairment, matched for age, body weight and, to the extent possible, for gender. The primary purpose of this study is to characterize the effect of renal impairment on the plasma pharmacokinetics of ALG-097558 following administration of multiple, twice daily (Q12H) oral (PO) doses.

ELIGIBILITY:
Inclusion Criteria for All Subjects:

1. Male and Female between 18 and 75 years old
2. Body Mass Index (BMI) 17.5 to 40.0 kg/m^2 and a total body weight >50 kg (110 lb)
3. Female subjects must either be not of childbearing potential or if they are a woman of childbearing potential, they are only eligible if they and any non-sterile, male sexual partners agree to use highly effective contraceptive therapy

Inclusion Criteria for Subjects with Normal Renal Function:

1. Good general health as defined by no clinically relevant abnormalities identified by Medical History and a vital signs, clinical laboratory and 12-lead electrocardiogram (ECG) assessment
2. Subjects must fit the demographic-matching criteria including body weight, age, and to the extent possible, gender
3. Normal renal function (estimated Glomerular Filtration Rate [eGFR] ≥90 mL/min) with no known or suspected renal impairment

Inclusion Criteria for Subjects with Impaired Renal Function:

1. Subject satisfies the eGFR criteria for renal impairment classification within 28 days of study drug administration
2. Any form of renal impairment except acute nephritic syndrome (subjects with history of previous nephritic syndrome but in remission can be included).
3. Stable concomitant medications for the management of an individual subject's medical history for at least 28 days prior to screening
4. Subjects must have a 12-lead ECG and vital signs assessment that meet the protocol criteria

Exclusion Criteria for All Subjects:

1. Subjects with any current or previous illness that, in the opinion of the Investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject or that could prevent, limit, or confound the protocol specified assessments or study results and interpretation
2. Subjects with a past history of cardiac arrhythmias, risk factors for Torsade de Pointes syndrome (e.g., hypokalemia, family history of long QT Syndrome) or history or clinical evidence at screening of significant (subjects with normal renal function) or unstable (subjects with renal impairment) cardiac disease etc.
3. Subjects with a history of clinically significant drug allergy
4. Subjects with a recent (within 1 year of randomization) history or current evidence of drug abuse or recreational drug use
5. Excessive use of alcohol defined as regular consumption of ≥14 units/ week for women and ≥21 units/week for men
6. Unwilling to abstain from alcohol use for 48 hours prior to start of the study through end of study follow up
7. Subjects with Hepatitis A, B, C, E or HIV-1/HIV-2 infection or acute infections such as SARS- CoV-2 infection
8. Subjects with alanine aminotransferase (ALT) or aspartate aminotransferase (AST) values >2x upper limit of normal (ULN)
9. Subjects with bilirubin (total, direct) >1.5x ULN (unless Gilbert's is suspected)
10. Positive pregnancy test; females must not be pregnant at enrollment

Exclusion Criteria for Subjects with Normal Renal Function:

1. Hemoglobin <10 g/dL

Exclusion Criteria for Subjects with Impaired Renal Function:

1. Participants requiring hemodialysis and/or peritoneal dialysis
2. Hemoglobin <9 g/dL

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-07-21 (Actual); Study Completion 2025-07-21 (Actual)

PRIMARY OUTCOMES:
Area under the concentration time curve [AUC] | Pre-dose (-0.75 hours) up to Day 8
  Pharmacokinetic parameters of ALG-097558 and metabolite ALG-097730 in plasma
Maximum plasma concentration [Cmax] | Pre-dose (-0.75 hours) up to Day 8
  Pharmacokinetic parameters of ALG-097558 and metabolite ALG-097730 in plasma
Minimum plasma concentration [Cmin] | Pre-dose (-0.75 hours) up to Day 8
  Pharmacokinetic parameters of ALG-097558 and metabolite ALG-097730 in plasma
C0 [predose] | Pre-dose (-0.75 hours) up to Day 8
  Pharmacokinetic parameters of ALG-097558 and metabolite ALG-097730 in plasma
Half-life [t1/2] | Pre-dose (-0.75 hours) up to Day 8
  Pharmacokinetic parameters of ALG-097558 and metabolite ALG-097730 in plasma
Time to maximum plasma concentration [Tmax] | Pre-dose (-0.75 hours) up to Day 8
  Pharmacokinetic parameters of ALG-097558 and metabolite ALG-097730 in plasma
Apparent Clearance (CL/F) | Pre-dose (-0.75 hours) up to Day 8
  Pharmacokinetic parameters of ALG-097558 and metabolite ALG-097730 in plasma
Apparent Volume of Distribution (V/F) | Pre-dose (-0.75 hours) up to Day 8
  Pharmacokinetic parameters of ALG-097558 and metabolite ALG-097730 in plasma
Total Amount of Drug Excreted in Urine (Ae) | Pre-dose (-0.75 hours) up to Day 8
  Pharmacokinetic parameters of ALG-097558 and metabolite ALG-097730 in urine
Renal Clearance (CLr) | Pre-dose (-0.75 hours) up to Day 8
  Pharmacokinetic parameters of ALG-097558 and metabolite ALG-097730 in urine

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 20 Days
  The number and severity of treatment emergent events in subjects with renal impairment and subjects with normal renal function as assessed by DAIDS v2.1 (July 2017)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Genesis Clinical Trials, Tampa, Florida